CLINICAL TRIAL: NCT02029287
Title: Remote Prevention and Treatment Based on Community Under the Guidance of Regional Central Hospital for Patients With Chronic Heart Failure
Brief Title: Hospital-Community-Family-Care Management Platform for Chronic Heart Failure
Acronym: HCF-CMP-CHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Gu (Other)
Collaborators: Science and Technology Department of Jiangsu Province (Unknown); Yangzhou Municipal Health Bureau (Unknown)
Responsible Party: Sponsor-Investigator, Xiang Gu, Professor of Cardiology, Director of Cardiovascular Medicine, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BL2013022
Record Dates: First submitted 2013-12-21; First posted 2014-01-07 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; telemedicine; health service platform

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects with CHF follow-up (Experimental): Subjects with Hospital-Community-Family-Care Management Platform online and those with the clinic follow up.In the program, participants were educated on the use of smart health-tracking devices and mobile application (APP) to collect and upload comprehensive data elements related to the risk of CHF self-care management. They were also instructed to send text messages, view notifications, and receive individualized guidance on the mobile APP. The general practitioners viewed index of each participant on mobile APP and provided primary care periodically, and cardiologists in regional central hospital offered remote guidance and management if necessary. Outcomes assessed included accomplishments of the program, usability and satisfaction, engagement with the intervention, and changes of heart failure-related health behaviors.
  Interventions: Other: Hospital-Community-Family-Care Management Platform Online; Other: Subjects with CHF via conventional clinic visit according to the latest relevant guidelines
- Subjects with CHF conventional clinic visit (Active Comparator): Subjects with standardized treatment according to latest guidelines via conventional visit.
  Interventions: Other: Subjects with CHF via conventional clinic visit according to the latest relevant guidelines

INTERVENTIONS:
Other: Hospital-Community-Family-Care Management Platform Online — Hospital-Community-Family-Care Management Platform Online: the remote monitoring service platform on line based on community and family for subjects with CHF under the guidance of the regional central hospital
  Other Names: Subjects with CHF follow-up
  Arms: Subjects with CHF follow-up
Other: Subjects with CHF via conventional clinic visit according to the latest relevant guidelines — Subjects with CHF via conventional clinic visit according to the latest relevant guidelines

SUMMARY:
The purpose of this study is to determine whether the Hospital-Community-Family-Care Management Platform for Chronic Heart Failure reduces the mortality, readmission rates and costs of the subjects with CHF.

DETAILED DESCRIPTION:
(1) Indication: Chronic Heart Failure. (2) Objectives: Primary objective is to evaluate the efficacy of the Hospital-Community-Family-Care Management Platform online compared with the regular clinic follow up in subjects with CHF (I-IV class by NYHA, of which class IV without strict bed rest).Secondary objectives is to assess the safety of the Management Platform online in subjects with CHF. (3) Study design: Prospective, randomized, controlled study with two follow up management groups: 1) the Hospital-Community-Family-Care Management Follow up Online; 2) the regular monthly clinic follow up. Study population: Totally 1000 male and female subjects with CHF (I-IV functional class according to NYHA classification). (4) Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing. (5) Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry. (6) Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources. (7) Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. (8) Duration of follow up: The total follow-up time shall be at least 12 months. (9) Safety Assessment: Safety of the study will be evaluated by the following assessments: 1) Subject and object examinations (during the follow up period and extending up to 2 week after the end of the study) consisting of a subject interview (including direct questioning about adverse events), physical examination, assessment of body weight, Electrocardiogram (ECG) and echocardiogram (UCG), Left ventricular ejection fraction (LVEF), assessed by echocardiography, The N-terminal prohormone of brain natriuretic peptide (NT-proBNP), a peptide hormone whose plasma concentration is inversely related to the severity of HF, NYHA functional status, assessed by subject interview, 6-minute walk distance (6MWD), Quality of life (QoL), assessed by the Minnesota Living with Heart Failure questionnaire (MLHFQ), a validated questionnaire assessing QoL in subjects with heart failure. 2) Evaluation of clinically relevant safety laboratory parameters, such as complete blood count, serum creatinine, electrolytes, and liver enzymes. Any Adverse Events (AE) or Serious Adverse Events (SAE) and its potential causal relationship with the study will be recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:to be considered eligible to participate in this study, a subject must meet the inclusion criteria listed below at the time of screening and randomization:

1. Male and female are aged 18 years old or over.
2. History of CHF for ≥3 months with NYHA functional class I-IV, of which class IV without strict bed rest.
3. Left ventricular ejection fraction (LVEF) ≤45% as assessed by echocardiogram. However, LVEF can be above 45% for patients with cardiac insufficiency caused by atrial fibrillation, valvular heart disease, hypertrophic cardiomyopathy and et al;
4. Treatment of CHF with stable and optimal pharmacological therapy according to Chinese guidelines for treatment of CHF. In general, optimal treatment will include a beta-blocker and an ACE inhibitor and/or an angiotensin receptor blocker, unless not tolerated. Medical therapy is defined as stable, if the subject has not started a new CHF drug class and the dose of drugs taken have not been changed during the 3 months prior to screening and randomization.
5. Ability to understand the requirements of the study and willingness to provide written informed consent (IC), and agreement to abide by the study restrictions and return for the required assessments.
6. Subjects are located in our coverage of the remote monitoring system.

Exclusion Criteria:To be eligible for entry into the study, the subject must not meet any of the exclusion criteria listed below at screening and randomization:

1. Some secondary cardiomyopathy: hyperthyroid heart disease and anemic heart disease, and et al;
2. A history of malignancy, and life expectancy is less than 1 year；
3. Severe primary hepatic and renal insufficiency (alanine aminotransferase≥100 u/L, serum creatinine >3.0mg/dL, serum albumin <2.5g/L);
4. Refusal to participate;
5. Unable to visit outpatient clinics periodically;
6. Ambulatory population;
7. Patients were considered inappropriate to participate by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-12; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year
  Number of subjects with all cause death

SECONDARY OUTCOMES:
Heart failure morbidity | one year
  number of subjects with heart failure - related visits

OTHER OUTCOMES:
heart failure worsening | one year
  Number of subjects requiring drug or dose changes to intensify concomitant therapy due to worsening of heart failure (HF).
Hospitalization rate | one year
  Hospitalization rate associated with heart failure
Average hospitalization time | one year
  Average hospitalization time associated with heart failure
Costs of medications | one year
  Costs of medications associated with heart failure
Usability of the HCF intervention for patients | 4 months
  it was assessed based on the Perceived Health Web Site Usability Questionnaire (PHWSUQ-12)
Changes of self-management | 4 months
  Lifestyle and health behaviors of participants were collected by interview
Engagement of the intervention | 4 months
  It was assessed objectively via daily Web portal log-ins and use of the mobile APP
Participants perceptions of intervention components | 4 months
  During the interview, qualitative method was used to examine participants perceptions of intervention components

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Gu, Docter, Principal Investigator — Department of cardiovascular medicine; Jianhua Shen, Docter, Principal Investigator — Department of cardiovascular medicine
Locations (1):
- Department of cardiovascular medicine,Northern Jiangsu Hospital, Yangzhou, Jiangsu, China